CLINICAL TRIAL: NCT06745973
Title: An Exploratory Clinical Study Evaluating EPI-003 Injection for the Treatment of Chronic Hepatitis B
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Epigenic Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPI-003-I01
Record Dates: First submitted 2024-12-09; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EPI-003 (Experimental)
  Interventions: Drug: EPI-003

INTERVENTIONS:
Drug: EPI-003 — Intravenous (IV) infusion.

SUMMARY:
This study is an open-label, 2-Part (Single Ascending Dose [Part 1] And Dose Expansion) study that will evaluate the safety of EPI-003 administered to patients with chronic infection with HBV (CHB). EPI-003 is a liver-targeted antiviral therapeutic for intravenous (IV) injection that is capable of precise epigenetic modifications of the HBV genome without causing mutations in the gene sequence itself.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 18 and 65 years of age, inclusive, at the time of signing the informed consent form;
2. Confirmed diagnosis of CHB;
3. Received a stable dose of NA therapy for ≥ 6 months prior to screening and plan to continue receiving the same dose for the duration of the study

Exclusion Criteria:

1. Confirmed diagnosis of liver cancer or cirrhosis;
2. Combination of other major diseases; 3 Pregnant or lactating females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs | From Baseline through to Day 28 postdose

SECONDARY OUTCOMES:
Evaluation of maximum observed concentration (Cmax) | From Baseline through to Day 28 postdose
Evaluation of maximum observed concentration (tmax) | From Baseline through to Day 28 postdose
Evaluation of terminal elimination half-life (t1/2) | From Baseline through to Day 28 postdose
HBsAg | From Baseline through to Day 365 postdose

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs). | From Baseline through to Day 365 postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No